CLINICAL TRIAL: NCT06479512
Title: Can Caval-aorta Index and Perfusion Index Predict Hypotension After Spinal Anaesthesia in Elderly Patients Undergoing Lower Extremity Surgery?
Brief Title: Caval-aorta Index and Perfusion Index on Predict Hypotension After Spinal Anaesthesia in Elderly
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Fatma Kavak Akelma, anesthesiology and reanimation associate professor, Ankara Yildirim Beyazıt University
Other Study IDs: spinal-induced hypotension
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia, Spinal
Keywords: spinal anesthesia; caval aorta index; perfusion index; orthopedic surgery; elderly patients
MeSH Terms: interventions — Perfusion Index

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with spinal induced hypotension: patients with hypotension after spinal anesthesia (SBP less than 90 mmHg, a decrease in SBP by more than 30% from the preoperative baseline value, or an MAP below 60 mmHg)
  Interventions: Device: ultrasonography to measure the index of the caval aorta and non-invasive pulse oximetry for perfusion index
- patients without spinal induced hypotension: patients without spinal induced hypotension
  Interventions: Device: ultrasonography to measure the index of the caval aorta and non-invasive pulse oximetry for perfusion index

INTERVENTIONS:
Device: ultrasonography to measure the index of the caval aorta and non-invasive pulse oximetry for perfusion index — Inferior vena cava and aortic diameter measurements will be made by ultrasonography and perfusion index determination using non-invasive pulse oximetry

SUMMARY:
The aim of our study was to predict hypotension by using caval aorta index and perfusion index in elderly patients who may develop hypotension after spinal anesthesia.

DETAILED DESCRIPTION:
The study will include 200 patients over 60 years of age who are planned to undergo elective lower extremity surgery in the supine position with spinal anaesthesia. This study is planned as a single-centre prospective observational study. All patients planned to be included in the study will be fasted according to the standard protocol. Age, height, body weight, body mass index, gender, type of surgery, systemic disease, preoperative heart rate (HR), noninvasive systolic (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP) and peripheral oxygen saturation (SpO₂) will be measured and noted in the waiting area before entering the operating room. For the initial perfusion index (PI) value, PI measurement will be taken 3 times at 5 minutes intervals with a probe to be attached to the same finger and the average will be recorded as the initial PI value. To measure the IVC diameter, the maximum internal AP diameter of the IVC will be measured in M-mode during expiration and the mean will be taken. The maximum internal AP diameter of the abdominal aorta will be measured during systole and the mean will be recorded as the aortic diameter.The study will be explained to all patients participating in the study and informed consent will be obtained from the patients. Routine preoperative preparations and monitoring of the patients admitted to the operating room will be performed. Spinal anaesthesia will be performed through L3-4 or L4-5 intervertebral spaces in the sitting position.Depending on the nature of the patient and the type of surgery, an appropriate dose of 0.5% hyperbaric bupivacaine will be injected intrathecally to provide adequate sensory block.The patient will be immediately placed in the supine position.The level of sensory blockade will be evaluated at the end of the appropriate time. heart rate, systolic, diastolic blood pressure, mean arterial pressure, oxygen saturation and PI will be recorded every 2 minutes for the first 15 minutes, then every 5 minutes until the 30th minute, then every 10 minutes until the 60th minute and at the end of the operation.Hypotension after spinal anaesthesia will be defined as SDB less than 90 mmHg, a fall in SDB by more than 30% from the preoperative baseline value or an OAB less than 60 mmHg.Patients will be divided into two groups as patients with and without hypotension after spinal anaesthesia. Demographic data (age, gender, comorbidity, etc.), caval-aorta index and PI will be analysed for differences between the groups.

The primary aim of the study was to evaluate the ability of caval-aorta index and PI to predict post-spinal hypotension in elderly patients between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology(ASA) I-II-III score
* Patients over 60 years
* Elective surgeries
* Surgeries in supine position

Exclusion Criteria:

* Patient refusal to participate in the study
* The patient will undergo emergency surgery
* Contraindication to spinal anaesthesia
* Planning unilateral spinal anaesthesia
* Failure of spinal anaesthesia
* Body mass index above 35kg/m2
* Presence of preoperative hypotension (SBP<90mmHg or MAP<60mmHg)
* The patient has valvular disease and arrhythmia impairing haemodynamics
* Presence of neuropsychiatric disorders that make communication difficult
* Presence of abdominal hernia

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients over 60 years of age who will undergo elective lower extremity surgery in supine position admitted to ankara city hospital
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
caval aorta index for predicting hypotension in the elderly | 1 hour
  to determine the threshold value for the caval aorta index in determining hypotension using logistic regression analysis

SECONDARY OUTCOMES:
perfusion index for predicting hypotension in the elderly | 1 hour
  to determine the threshold value for the perfusion index in determining hypotension using logistic regression analysis
inferior vena cava diameter for predicting hypotension in the elderly | 1 hour
  to determine the threshold value for the inferior vena cava diameter in determining hypotension using logistic regression analysis
abdominal aort diameter for predicting hypotension in the elderly | 1 hour
  To determine the effect of abdominal aort diameter on the prediction of hypotension using logistic regression analysis.
systolic blood pressure | 1 hour
  recorded preoperatively and in the operating room every 2 minutes for the first 15 minutes, then every 5 minutes until the 30th minute, then every 10 minutes until the 60th minute and at the end of the operation
diastolic blood pressure | 1 hour
  recorded preoperatively and in the operating room every 2 minutes for the first 15 minutes, then every 5 minutes until the 30th minute, then every 10 minutes until the 60th minute and at the end of the operation
mean arterial pressure | 1 hour
  recorded preoperatively and in the operating room every 2 minutes for the first 15 minutes, then every 5 minutes until the 30th minute, then every 10 minutes until the 60th minute and at the end of the operation
hearth rate | 1 hour
  recorded preoperatively and in the operating room every 2 minutes for the first 15 minutes, then every 5 minutes until the 30th minute, then every 10 minutes until the 60th minute and at the end of the operation
oxygen saturation | 1 hour
  recorded every 2 minutes for the first 15 minutes, then every 5 minutes until the 30th minute, then every 10 minutes until the 60th minute and at the end of the operation
bromage scale motor blocage score | 1 hour
  bromage scale score is a score between 0 and 3. bromage 0 means full movement of the leg and knee, bromage 3 means full motor blockade of the legs. the time to reach bromage 3 will be recorded
T10 dermatome | 1 hour
  time to reach T10 dermatome level
dermatomal level | 1 hour
  the highest dermatome level achieved with spinal anesthesia
use ephedrine | 1 hour
  dose of ephedrine used

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Ankara, Çankaya, Turkey, 06800, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No